CLINICAL TRIAL: NCT04158037
Title: Don't Go There: A Geospatial mHealth App for Gambling Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical difficulties with the mHealth app development
Sponsor: St. Louis University (Other)
Collaborators: National Center for Responsible Gaming (Other)
Responsible Party: Principal Investigator, Jeremiah Weinstock, Associate Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30494
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Gambling Disorder
Keywords: mHealth App
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth App (Experimental): Participants will receive the gambling disorder mHealth app.
  Interventions: Behavioral: mHealth App
- Wait List Control (No Intervention): Participant will be placed on a wait list for 12 weeks, after which they will be offered the gambling disorder mHealth app.

INTERVENTIONS:
Behavioral: mHealth App — The app uses smartphones' global positioning software (GPS) that recognizes a user's location to within 15 feet. The app will construct a customizable geofence (e.g., 3 miles) around a gambler's favored gambling venue (e.g., casino, gas station). If the individual crosses the fence boundary his or her phone will raise the alarm with a personalized motivational message.
  Arms: mHealth App

SUMMARY:
The goal of this project is to develop and to test the efficacy of a novel mHealth app for gambling disorder. The app capitalizes on smartphones' global positioning software (GPS) that recognizes a user's location to within 15 feet. Users will receive an alert of this go near a gambling venue. The project will conduct a 12-week pilot randomized clinical trial to test the short-term efficacy of the app with gambling disorder individuals.

ELIGIBILITY:
Inclusion Criteria:

* Currently meets DSM-5 criteria for gambling disorder
* At least 4 non-online gambling episodes in past 60 days
* Wagering at least $100 total over past 60 days
* Willingness to accept random assignment
* English speaking
* Android phone user

Exclusion Criteria:

* Age <18 years old
* Severely disruptive behavior
* Serious uncontrolled psychiatric behavior that requires acute psychiatric care
* Decline permission to collect zero permission data from smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
App usage (feasibility) | From baseline to post-treatment (12 weeks)
  Number of days the app is active on a user's smartphone. Days can range from 0 to 84.
Patient satisfaction with the gambling app | From baseline to post-treatment (12 weeks)
  Investigator derived patient satisfaction self-report questionnaire. Five items, using a 7-point Likert scale from very dissatisfied (1) to very satisfied (7). Higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Gambling behavior via Timeline Followback (Weinstock, Whelan, & Meyers, 2004) | From baseline to post-treatment (12 weeks)
  Self-report gambling frequency and intensity as assessed by the Gambling Timeline Followback - a retrospective self-report calendar. Gambling frequency can range from 0 to 84; gambling intensity is measured in $ and time (hours). Dollars wagered can range from $0 to unlimited $. Time is measured in hours and can range from 0 to >1,000 hours. Higher scores indicate a worse outcome.
Gambling-related harms (Browne et al., 2018) | From baseline to post-treatment (12 weeks)
  Self-reported gambling harms as assessed by the 72-item Gambling-Related Harms Questionnaire (yes/no responses). Scores range from 0 to 72. Higher scores indicate a worse outcome.
Quality of Life Inventory (Frisch et al., 1994). A self-reported quality of life measure assessing 17 domains of life for importance and satisfaction. | From baseline to post-treatment (12 weeks)
  Self-report quality of life questionnaire. Participants rate 17 domains on importance (range not at all important [0] to extremely important [2]). The 17 domains are then rated on how satisfied the individual is regards to his or her life (-3 [very dissatisfied] to 3 [very dissatisfied]). A total score is then generated by summing the product of importance multiplied by satisfaction. Scores range from 0 to 102. Higher scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremiah Weinstock, PhD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No